CLINICAL TRIAL: NCT03605550
Title: A Phase 1b Study of PTC596 in Children With Newly Diagnosed Diffuse Intrinsic Pontine Glioma and High Grade Glioma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CONNECT1702; 5R01FD006352-03 (FDA)
Record Dates: First submitted 2018-07-20; First posted 2018-07-30 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: High Grade Glioma; Diffuse Intrinsic Pontine Glioma
Keywords: DIPG; High Grade Glioma
MeSH Terms: conditions — Glioma; Diffuse Intrinsic Pontine Glioma | interventions — PTC596; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (PTC596) (Experimental): PTC596 administered orally twice weekly (M/Th or T/F schedule) concomitantly with RT for 6 -7 weeks. Each subsequent cycle is defined as 28 days. Post RT patients will continue to receive PTC596 twice weekly for up to 26 cycles at RP2D of 200mg/m2 with a maximum dose capped at 400mg for patients with BSA ≥2.0
  Interventions: Drug: PTC596; Radiation: Radiotherapy

INTERVENTIONS:
Drug: PTC596 — Oral tablets
Radiation: Radiotherapy — Cycle1

SUMMARY:
The goal of this study is to evaluate the safety of the study drug PTC596 (Unesbulin) taken in combination with radiotherapy (RT) when given to pediatric patients newly diagnosed with High-Grade Glioma (HGG) including diffuse intrinsic pontine glioma (DIPG).

The main aims of the study are to:

* Find the safe dose of the study drug PTC596that can be given without causing serious side effects.
* Find out the amount of drug that enters blood (in all patients) and tumor (in patients who receive drug prior to a planned surgery for removal of their brain tumor)

During the first cycle (6-7weeks), patients will receive drug orally twice a week in combination with daily RT. During subsequent cycles (4 weeks each), they will receive only the study drug orally twice a week.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
This study consists of 3 parts:

1. The Phase I (Parts A and C), dose-finding component of the trial, to estimate the maximum tolerated dose (MTD) or recommended phase II dose (RP2D) of PTC596 in combination with RT followed by maintenance therapy with PTC596, in children with newly-diagnosed DIPG and HGG.

   Once the RP2D has been determined,
2. An early efficacy expansion cohort of up to 17 patients at the RP2D (Part C expansion, and Part D)
3. A surgical cohort (part B) of 12 patients with newly diagnosed DIPG who are amenable to undergo biopsy or HGG for whom a second surgical resection is warranted

For patients on cohorts A, C and D, PTC596 will be given orally twice weekly for 6-7 weeks along with daily RT for the first cycle. In subsequent cycles (4 weeks each), all patients will continue with maintenance therapy which will begin immediately after completion of RT for up to 26 cycles (2 years).

For the surgical cohort, patients will be treated with 2 doses of PTC596, on days 1 and 4 prior to biopsy or re-resection; the second dose of PTC596 should ideally be administered 3-6 hrs before surgery. The surgical cycle will end when patients begin RT which should take place at least two weeks after the date of surgery and may restart PTC596 (twice weekly) after starting RT. Following completion of RT, patients will immediately start maintenance therapy with twice weekly PTC596 for up to 26 cycles.

Primary Objectives Parts A, C

* To determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of PTC596 given concurrently with radiation in newly-diagnosed patients with DIPG or HGG (Parts A and C)
* To determine the toxicities of PTC596 given concurrently with RT and during maintenance therapy (Parts A, C).
* To characterize the pharmacokinetics of PTC596 given as a capsule and as a tablet in children with newly diagnosed DIPG or HGG when given concurrently with RT and during maintenance (Parts A, C).

Primary Objectives Surgical Cohort -Part B

* To test the ability of PTC596 to inhibit BMI-1 activity in tumor and PBMCs
* To characterize the pharmacokinetics of PTC596 in plasma, cerebrospinal fluid (CSF), and tumor tissue

Secondary Objectives

* To evaluate the overall survival (OS) for newly-diagnosed patients with DIPG treated with PTC596 and compare to historical controls.
* To estimate the progression-free survival (PFS) distribution for newly-diagnosed patients with HGG ttreated with PTC596 and compare to historical controls
* To determine the effects of BMI-1 modulation in DIPG and HGG on BMI-1 levels, H2A monoubiquitination, cell proliferation, cell death, gene regulation, through gene expression profiling and epigenetic studies such as RNA sequencing and ChIP-Seq within the confines of a Phase I study.
* Correlate pre-treatment and post-treatment concentrations of potential biomarkers in biological specimens (e.g., blood and tissue) with response/toxicity, PFS, OS within the confines of a phase I study.
* To examine H3F3A, HIST1H3B (H3.3 and H3.1 genes), ATRX, and DAXX mutations and examine the effects of these alterations using targeted gene, exome, RNA sequencing and methylation arrays of targeted genomic regions in DIPG and HGG.
* To assess the health-related quality-of-life of patients by parent report, and when possible, patient report at key points in therapy using the patient reported outcomes measurement information system (PROMIS) survey.
* To explore tumor volumetric measurements on MRI and correlate with 2-dimensional measurements and compare response criteria.
* To correlate early measures of tumor response (volumetric and 2-dimensional measurements with overall survival.

ELIGIBILITY:
Inclusion Criteria:

Age: Patients must be ≥12 months and ≤ 21 years of age at the time of study enrollment.

Diagnosis: Patients with newly-diagnosed diffuse intrinsic pontine gliomas (DIPGs), defined as tumors with a pontine epicenter and diffuse involvement of at least 2/3 of the pons, are eligible without histologic confirmation.

Patients with brainstem tumors that do not meet radiographic criteria or are not considered to be typical diffuse intrinsic pontine gliomas will be eligible if the tumors are biopsied and proven to be high-grade gliomas (such as anaplastic astrocytoma, glioblastoma, H3K27-mutant diffuse midline glioma) or diffuse astrocytoma.

Patients with newly-diagnosed non-brainstem high-grade glioma (HGG) are eligible.

Patients must have had histologically verified high-grade glioma such as anaplastic astrocytoma, glioblastoma, H3 K27 mutant diffuse midline glioma etc.

Patients eligible for the surgical stratum include patients with:

1. Newly-diagnosed DIPG who are amenable to undergo biopsy at the recommendation of their treating physician
2. Newly-diagnosed HGG for whom a second surgical resection is warranted for further debulking or to achieve a near-total or gross total resection after initial diagnosis has been made but prior to start of therapy.

   Disease Status: Patients with disseminated DIPG or HGG are not eligible, and MRI of spine must be performed if disseminated disease is suspected clinically by the treating physician.

   Performance Level: Karnofsky ≥ 50 for patients > 16 years of age and Lansky ≥ 50 for patients ≤ 16 years of age. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.

   Neurologic Status: Patients must be able to swallow oral medications to be eligible for study enrollment.

   Patients enrolling on Part A (phase I, capsule formulation) must be able to swallow whole capsules.

   Prior Therapy: Patients must not have received any prior anticancer therapy. Prior dexamethasone and/or surgery are permissible.

   Organ Function Requirements:

   Adequate Bone Marrow Function Defined as:

   • Peripheral absolute neutrophil count (ANC) ≥ 1000/mm3

   • Platelet count ≥ 100,000/mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)

   • Hemoglobin >8 g/dL (may be transfused).

   Adequate Renal Function Defined as:

   • Creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73 m2 or

   • A serum creatinine based on age/gender as follows:
   * 1 to < 2 years: 0.6 (Male) 0.6 (Female)
   * 2 to < 6 years: 0.8 (Male) 0.8 (Female)
   * 6 to < 10 years: 1 (Male) 1 (Female)
   * 10 to < 13 years: 1.2 (Male) 1.2 (Female)
   * 13 to < 16 years: 1.5 (Male) 1.4 (Female)

     * 16 years: 1.7 (Male) 1.4 (Female)

   Adequate Liver Function Defined as:

   • Total bilirubin must be ≤ 1.5 times institutional upper limit of normal for age

   • AST(SGOT)/ALT(SGPT) < 3 times institutional upper limit of normal

   • Serum albumin ≥ 2g/dL

   Adequate Cardiac Function Defined As:

   - Ejection fraction of ≥ 55% by echocardiogram.

   - QTc ≤ 480 msec.

   Adequate Pulmonary Function Defined as

   - No evidence of dyspnea at rest, and a pulse oximetry > 94% in room air if there is clinical indication for determination

   Adequate Neurologic Function Defined as:

   - Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled.

   Informed Consent: All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.

   Exclusion Criteria:

   Diagnosis: patients with a diagnosis of oligodendroglioma or oligoastrocytoma are not eligible. Patients with juvenile pilocytic astrocytoma, are not eligible.

   Patients with non-brainstem diffuse astrocytoma (grade 2) are not eligible for the HGG stratum of the study.

   Pregnancy or breast-feeding: Pregnant or breast-feeding women will not be entered on this study due to known or unknown risks of fetal and teratogenic adverse events as seen in animal/human studies. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.

   Patients of childbearing or child fathering potential must agree to use adequate contraceptive methods (hormonal or barrier method of birth control; abstinence) while being treated on this study and for 3 months after completing therapy. Note: The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.

   Concomitant Medications
   * Corticosteroids: Patients receiving corticosteroids are eligible. The use of corticosteroids must be reported.
   * Investigational Drugs: Patients who are currently receiving another investigational drug are not eligible.
   * Anti-cancer Agents: Patients who are currently receiving other anti-cancer agents are not eligible.
   * Anticonvulsants: Patients who are receiving enzyme inducing anticonvulsants as listed in appendix II, are not eligible
   * Patients who are receiving rifampin are not eligible.
   * Patients who are receiving medications known to prolong QTc interval as listed in appendix III are not eligible.
   * Patients who are receiving duloxetine, alosetron or theophylline (CYP1A2 inhibitors) are not eligible
   * Patients on beta-blockers are not eligible
   * Selective serotonin reuptake inhibitors (SSRIs) such as citalopram (Celexa), escitalopram (Lexapro), Fluoxetine (Prozac), fluvoxamine (Luvox), paroxetine (Paxil), sertraline (Zoloft) should be used with caution but are not contraindicated.
   * Anticoagulants: patients who are receiving therapeutic anticoagulants including warfarin, low-molecular weight heparin are not eligible

   Nasogastric or G tube administration of PTC596 is not permissible.

   Infection: Patients who have an uncontrolled infection are not eligible.

   Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study are not eligible.

   Patients with evidence of bowel obstruction, malabsorption, or other contraindication to oral medication are not eligible.

   Patients with GI disease or other condition that could affect absorption or predispose subject to gastrointestinal ulceration are not eligible.

   Patients with an active peptic ulcer disease or inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis are not eligible.

   Patients with serious non-healing wounds, ulcers, or bone fractures are not eligible.

   Patients with moderate to severe pulmonary problems generally defined by need for medical intervention (e.g., oxygen, medications) and/or limiting activities of daily living (generally CTCAE Grade 2 or higher) or shortness of breath with limited exertion are not eligible. Pulmonary conditions include (but are not limited to) COPD, asthma, and hemi-pneumectomy.

   Patients with malignancy related to HIV or solid organ transplant: known history of HIV, HBV surface antigen positivity or positive HCV antibody are not eligible. Viral testing is not required unless clinically indicated in patients without a known history.

   Patient with prior or ongoing clinically significant illness, medical or psychiatric condition, medical history, physical findings, ECG findings, or laboratory abnormality that, in the investigator's opinion, could affect the safety of the subject, or alter the absorption, distribution, metabolism, or excretion of the study drugs, or could impair the assessment of study results are not eligible.

   Patients with any prior solid organ transplant are not eligible

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Establish MTD and RP2D of PTC596 | At the end of Cycle 1 (42-49 days)
  To determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of PTC596 given concurrently with radiation in newly-diagnosed patients with DIPG or HGG (Parts A and C)
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | From Day 1 of treatment through 30 days following end of protocol treatment
  To determine the toxicities of PTC596 given concurrently with radiotherapy and during maintenance therapy (Parts A, C) in newly diagnosed HGG and DIPG patients treated with PTC596 by calculating the number of participants with, as well as frequency and severity of, PTC596-related Adverse Events as assessed by CTCAE v5.0.
Maximum Plasma Concentration [Cmax] of PTC596 (A, B, C, D) | Days1 through 29
  To characterize the plasma pharmacokinetics of PTC596 in children with newly-diagnosed DIPG or HGG when given concurrently with radiotherapy and during maintenance (Parts A, C, D) by measuring the Maximum Concentration [Cmax] and Area Under the Curve (AUC) of PTC596 in plasma
Tumor Concentration of PTC596 (B) | Day 4 of surgical cycle
  To characterize the pharmacokinetics of PTC596 in tumor tissue of children with newly-diagnosed DIPG and HGG who are treated with PTC596 before undergoing a second resection
Protein levels of BMI1 in tumor | Day 4 of surgical cycle
  To test the ability of PTC596 to inhibit BMI-1 activity and downstream effectors by measuring protein levels in tumor and peripheral blood mononuclear cells (PBMCs) of children with newly-diagnosed HGG and DIPG who are treated with PTC596 before undergoing a second resection

SECONDARY OUTCOMES:
Evaluate Overall survival | From date of treatment until date of death due to any cause or date of last follow-up, assessed up to 60 months
  To estimate the overall survival distribution for newly-diagnosed patients with high-grade glioma treated with PTC596 during radiotherapy followed by PTC596 and compare to historical controls
Evaluate Progression Free survival | From date of treatment until date of progressive disease or death due to any cause or date of last follow-up, assessed up to 60 months
  To estimate the progression-free survival distribution for newly-diagnosed patients with high-grade glioma treated with PTC596 during radiotherapy followed by PTC596 and compare to historical controls

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Fouladi, MD, Study Chair — Nationwide Children's Hospital; Patricia Baxter, MD, Study Chair — Baylor College of Medicine; Margot Lazow, MD, Study Chair — Nationwide Children's Hospital
Locations (10):
- United States (10):
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided
IPD would only be shared following publication of the study.